CLINICAL TRIAL: NCT03848585
Title: Improvement of Medicine Adherence and the Following Positive Effects on Transplants in Patients After Organ Transplantation With Pilloxa's Electronic Pillbox
Brief Title: Medicine Adherence and Effects on Transplants With Pilloxa's Electronic Pillbox
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Pilloxa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0001
Record Dates: First submitted 2019-02-15; First posted 2019-02-21 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Kidney Transplant; Complications; Liver Transplant; Complications
Keywords: Immunosuppressants; Treatment adherence
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The analysis is blinded. The statistician will not have access to the affiliation of the users until the statistical analysis of the study data is finalised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilloxa Pillbox (Experimental)
  Interventions: Device: Pilloxa Pillbox
- Non active Pilloxa Pillbox (Sham Comparator)
  Interventions: Other: Non active Pilloxa Pillbox

INTERVENTIONS:
Device: Pilloxa Pillbox — A Pilloxa Pillbox is used for the prescribed immunosuppressants.
  Arms: Pilloxa Pillbox
Other: Non active Pilloxa Pillbox — A Pilloxa Pillbox with reminders disabled and without active mobile application is used for the prescribed immunosuppressants.
  Arms: Non active Pilloxa Pillbox

SUMMARY:
Poor adherence to medication among patients with chronic diseases is a major problem. A patient group where the adherence to prescribed medications is extremely important are organ transplanted patients. It is well established that lack of adherence to immunosuppressive medication drastically increases the risk of rejection reactions, graft loss and deaths.

Pilloxa is a device meant to help users manage medication and support adherence to medication. This study evaluates if Pilloxa improves adherence to treatment for transplanted patient compared with conventional management. Patients who have received a transplanted kidney or liver will be studied.

Pilloxa is a system comprising of: a box with 14 separate containers to temporarily store tablets/capsules in and that can be open by 14 independent lids, a smartphone application and cloud based servers. The pillbox will at given times detect if pills are present in the different compartments and can connect, send and receive information to/from mobile application and the cloud.

ELIGIBILITY:
Inclusion Criteria:

* Patient had an organ (liver or kidney) transplanted.
* Patient who wishes to participate in the study and who is able to understand, read, write and give written informed consent in the Swedish or English language. For persons under the age of 18, the guardians must understand, read, write and give written informed consent in the Swedish or English language.
* Ongoing daily immunosuppressive medication that is expected to continue during the study period.
* Handles medication by herself or, in the case of children, that medication is handled by the guardian.
* The patients doses of immunosuppressants fits into the chambers of the product.
* The patient's medicine ordination is not expected to change more often than once weekly.
* Owns and uses a compatible smartphone, option for underage children that guardians hold a compatible smartphone.

Exclusion Criteria:

* Suffers from dementia, neurological disease or other cognitive impairment which causes problems in understanding instructions or managing medication independently.
* Physical inability to use the product as intended.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Adherence to medication | During 6 months
  The proportion of days with adherence to medication for each patient. Adherence is defined as taking drugs within the interval within 120.0 minutes before to 120.0 minutes after each prescribed dose.

SECONDARY OUTCOMES:
Organ rejection | During 6 months
  The incidence of biopsy verified acute and chronic rejections between the intervention and control groups will be studied.
Concentration of Tacrolimus | Clinical routine sampling during 6 months
  The patients trough levels of tacrolimus will be compared between the groups. Optimal trough target zone is defined according to the recommended levels. Standard deviation of the variations of trough levels in each patient will also be compared between the groups.
Graft Function - Creatinine | Clinical routine sampling during 6 months
  Study the Creatinine (both kidney and liver) levels between the intervention and control group.
Graft Function - eGFR | Clinical routine sampling during 6 months
  Study the Estimated glomerular filtration rate (eGFR, kidney transplantation) between the intervention and control group.
Graft Function - Bilirubin | Clinical routine sampling during 6 months
  Study the Bilirubin levels between the intervention and control group.
Graft Function - ALAT | Clinical routine sampling during 6 months
  Study the Alanine aminotransferase (ALAT) levels between the intervention and control group.
Graft Function - ASAT | Clinical routine sampling during 6 months
  Study the Aspartate aminotransferase (ASAT) levels between the intervention and control group.
Graft Function - INR | Clinical routine sampling during 6 months
  Study the International normalized ratio (INR) between the intervention and control group.
Graft Function - Gamma-GT | Clinical routine sampling during 6 months
  Study the Gamma-glutamyl transferase (Gamma-GT) levels between the intervention and control group.
Graft Function - ALP | Clinical routine sampling during 6 months
  Study the Alkaline phosphatase (ALP, liver transplantation) levels between the intervention and control group.
Graft survival and patient survival | During 6 months
  Definition of graft loss:
  Liver: Re-transplantation or death Kidney: Patient back on dialysis or death.
Quality of Life | At 6 months compared to baseline
  The numbers of acute re-admissions for intervention will be studied and compared between the groups.
  Changes in scoring generated using Rand-36 evaluation of medical outcomes pre and after the study period will be evaluated between the groups.
Serious Adverse Events and Adverse Events | During 6 months
User-friendliness | At 6 months
  The user-friendliness of the pillbox will be compared between the groups with surveys designed by Pilloxa.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Söderdahl, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Patient Area Transplantation, Karolinska University Hospital, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829